CLINICAL TRIAL: NCT05046171
Title: Decreasing Polypharmacy in Older Adults With Curable Cancers: a Pilot Cluster-randomized Trial
Brief Title: Decreasing Polypharmacy in Older Adults With Curable Cancers Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erika Ramsdale, Associate Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMLT19186; K08CA248721 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-09-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Older Adults; Cancer receiving chemotherapy; Polypharmacy
MeSH Terms: conditions — Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Pharmacist-led deprescribing intervention (Experimental): Pharmacists will complete a comprehensive medication assessment with the participant via telemedicine and discuss tailored recommendations for discontinuations of potentially inappropriate medications. The pharmacist will document the evaluation and recommendations and communicate to the participant and care team members. The pharmacist will telephone each participant at least one time after the initial intervention to assess adherence to instructions and recommendations, and to assess any symptoms potentially related to medication discontinuation.
  Interventions: Other: Pharmacist-led deprescribing
- Arm 2: Patient education brochure (Active Comparator): Participants will receive a brochure discussing medication appropriateness and deprescribing in general terms
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Pharmacist-led deprescribing — A pharmacist recruited onto the study will review the patient's current medication list and develop a list of targeted recommendations for deprescribing using the 3-step potentially inappropriate medications identification method.
  Arms: Arm 1: Pharmacist-led deprescribing intervention
Other: Patient education — Subjects receive a written pamphlet about deprescribing.
  Arms: Arm 2: Patient education brochure

SUMMARY:
This is a single-site cluster-randomized trial to assess efficacy and implementation outcomes of deprescribing interventions in 72 older adults with polypharmacy (PP) and curable cancers initiating chemotherapy. Oncologists (as the cluster) will enroll 6 patients each and will be randomized to either a pharmacist-led deprescribing intervention or patient education intervention. Initial focus groups with oncologists, nurses, pharmacists, primary care physicians, and patients will provide data for initial adaptations to the pharmacist-led intervention arm, and 8 patients will be enrolled as a pre-trial cohort to further refine and adapt the pharmacist-led intervention.

DETAILED DESCRIPTION:
Polypharmacy (PP), or the concurrent use of multiple medications, affects up to 92% of older adults with cancer. It has been associated with adverse outcomes in these patients including poor adherence to and tolerance of cancer therapy, decrease in physical functioning, unplanned hospitalizations, falls, increased symptoms, and lower survival. "Deprescribing," or the planned discontinuation of medications which may be potentially unsafe or inappropriate, is an intervention strategy which has the potential to decrease PP and improve outcomes. Deprescribing has not been studied in older adults with cancer receiving chemotherapy. The proposed study will adapt and refine potentially scalable deprescribing interventions, investigate the effects of deprescribing interventions on relative dose intensity and other adverse outcomes in older adults undergoing curative-intent chemotherapy, and identify barriers and facilitators of deprescribing interventions for patients, oncologists, and pharmacists. Focus groups and interviews with pharmacists, oncologists, nurses, primary care providers, and patient advocates will allow initial adaptation of the proposed interventions. A "pre-pilot" cohort of 8 patients with PP and cancer planned to receive curative-intent chemotherapy will undergo a pharmacist-led deprescribing intervention with additional iterative adaptations. Then, 72 patients will be allocated to a pharmacist-led deprescribing intervention versus patient education intervention in a cluster-randomized trial of 12 oncologist clusters.

ELIGIBILITY:
Inclusion Criteria:

* Be age ≥65 years;
* Have a diagnosis of malignancy including aggressive lymphoma or cancers of the breast, gastrointestinal system, genitourinary system, or lung;
* Be initiating chemotherapy, alone or in combination with other systemic antineoplastic agents, (for a period of at least 3 months) within 4 weeks of enrollment;
* Screen positive for polypharmacy (>10 medications) or potentially inappropriate medications
* Be able to read and write English;
* Be able to give informed consent, as determined by the primary oncologist, or has a legally authorized representative to sign consent in the case of cognitive impairment.

Exclusion Criteria:

* Be planned to receive a cancer treatment regimen that does not include standard cytotoxic chemotherapy (e.g., only targeted therapies, hormonal therapies, monoclonal antibody therapies, immunotherapy, etc.),
* Have surgery or radiation without concurrent chemotherapy planned within 3 months of consent,
* Have a planned referral to the geriatric oncology clinic (SOCARE) within one month of treatment initiation,
* Lack decisional capacity, if a legally authorized representative is not available to sign consent and participate in study visits and follow-up phone calls.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change between arms in Relative dose intensity (RDI) of chemotherapy | 12 Weeks
  Relative dose intensity (RDI) of chemotherapy, based upon standard dosing from National Comprehensive Cancer Network guidelines or similar reference. RDI assesses the proportion of planned therapy that the patient receives within 12 weeks of initiation of chemotherapy.

SECONDARY OUTCOMES:
Change between arms in Changes in functional status | 12 Weeks
  Changes in functional status, based on Instrumental Activities of Daily Living (IADL)
Change between arms in Changes in functional status | 12 Weeks
  Changes in functional status, based on Activities of Daily Living (ADL)
Change between arms in Grade 3-5 chemotherapy toxicity | 12 Weeks
  Grade 3-5 chemotherapy toxicity based on Common Terminology Criteria for Adverse Events (CTCAE) v.5
Hospitalizations | 12 Weeks
  assessed as ≥1 or 0
Patient-reported falls | 12 Weeks
  assessed as ≥1 or 0
Patient-reported symptoms | 12 Weeks
  Patient-reported symptoms, assessed by selected elements of the NCI Patient Reported Outcomes CTCAE (PRO-CTCAE, 10-20 items).

OTHER OUTCOMES:
Change between arms in implementation | 2 years
  Barriers and facilitators of intervention (implementation outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Ramsdale E, Mohamed M, Holmes HM, Zubkoff L, Bauer J, Norton SA, Mohile S. Decreasing polypharmacy in older adults with cancer: A pilot cluster-randomized trial protocol. J Geriatr Oncol. 2024 Mar;15(2):101687. doi: 10.1016/j.jgo.2023.101687. Epub 2024 Feb 1. PMID 38302299
- [Derived] Ramsdale E, Malhotra A, Holmes HM, Zubkoff L, Wang J, Mohile S, Norton SA, Duberstein PR. Emotional barriers and facilitators of deprescribing for older adults with cancer and polypharmacy: a qualitative study. Support Care Cancer. 2023 Oct 17;31(12):636. doi: 10.1007/s00520-023-08084-9. PMID 37847423